CLINICAL TRIAL: NCT03412305
Title: Effect of Antibiotic Prophylaxis in Dental Implant Surgery - a Multicenter Placebo-controlled Double-blinded Randomized Clinical Trial
Brief Title: The Effect of Antibiotic Prophylaxis Associated With Dental Implant Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Malmö University (Other)
Responsible Party: Principal Investigator, Bengt Götrick, associate professor, Malmö University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AB-IMP
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Infection Control; Antibiotic Prophylaxis
Keywords: Dental implants, antibiotic prophylaxis
MeSH Terms: interventions — Amoxicillin

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The tablets corresponding to each patient is packed in a container by the manufacturer of the trial drug. Each drug container is labeled by a code number (1-1000) and the contents of the containers are distributed according to a randomization list with block size 6. Randomization is thus carried out by the manufacturer, independent of investigator and participating clinicians.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amoxicillin oral tablets (Active Comparator): 2 g amoxicillin tablets orally 1 hour before implant placement
  Interventions: Drug: Amoxicillin
- Placebo (Placebo Comparator): Placebo tablets orally 1 hour before implant placement
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Amoxicillin — Antibiotic prophylaxis consisting of 4 amoxicillin tablets, totally 2 g, orally 1 hour before implant placement
  Other Names: Amoxicillin oral tablets
  Arms: Amoxicillin oral tablets
Other: Placebo — Placebo consisting of 4 tablets, orally 1 hour before implant placement
  Other Names: Placebo oral tablets (for Amoxicillin)
  Arms: Placebo

SUMMARY:
The overall aim of the study is to investigate whether routine administration of antibiotic prophylaxis 1 hour prior to implant surgery may prevent postoperative infection and implant loss in healthy or substantially healthy patients (ASA Class 1 and Class 2).

DETAILED DESCRIPTION:
The prevalence of bacteria resistant to antibiotics is increasing and there is a correlation between high consumption of antibiotics and high incidence of antibiotic resistance. It is therefore important to reduce the prescription of antibiotics. Antibiotics in dental care are used to treat oral infections as well as to prevent infections associated with surgical procedures. An example of the latter is antibiotic prophylaxis associated with dental implant surgery in order to reduce the risk of postoperative infection that can lead to loss of implant.The study will be conducted as a multicenter placebo-controlled randomized clinical trial. Eligible patients will be asked for participation and those who leave oral and written information will be included in the study. Patients included will be allocated to either active treatment (antibiotic prophylaxis) or placebo. Both clinicians and patients will be blinded to group affiliation. A total of 10 clinicians in 8 centers in the south of Sweden have agreed to participate and each clinicians will be allowed to use the implants and routines that they usually work with.

Specific aims of the study are to test the following hypotheses:

1. There is no difference in proportion of patients with early implant losses in patients receiving 2 g of amoxicillin preoperatively and patients receiving identical placebo tablets.
2. There is no difference in proportion of patients with early infections between patients receiving 2 g of amoxicillin preoperatively and patients receiving identical placebo tablets.
3. There is no difference in infections (within 3-6 months postoperatively) between patients receiving 2 g of amoxicillin preoperatively and patients receiving identical placebo tablets.

If it appears that antibiotic prophylaxis does not lead to any risk reduction, this result may provide a basis for guidelines rejecting antibiotic prophylaxis in dental implant surgery.

ELIGIBILITY:
Inclusion Criteria:

* Requirement for dental implant placement
* Over 18 years of age

Exclusion Criteria:

* Immunosuppressed or immunocompromised
* Affected by not controlled diabetes
* Serious or severe systemic disease (ASA classification > 2)
* Previous radiotherapy to the head or neck area
* Ongoing acute or chronic infection in the oral cavity
* Ongoing treatment with antibiotics
* Hypersensitivity to penicillin
* Previous or ongoing treatment with bisphosphonates
* In need of major bone augmentation
* Planned direct loading or early loading (within 2 weeks) of the implant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Implant failure | 3-6 months after implant placement
  Early implant mobility and/or infection, which requires the implant to be removed.

SECONDARY OUTCOMES:
Postoperative infection | 7-14 days after implant placement
  Presence of swelling, redness, pus, pain and wound dehiscence
Infection | 3-6 months after implant placement
  Presence of any type of infection such as abscess, fistula

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Götrick, Principal Investigator — Malmö University
Locations (1):
- Malmö university, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Momand P, Becktor JP, Naimi-Akbar A, Tobin G, Gotrick B. Effect of antibiotic prophylaxis in dental implant surgery: A multicenter placebo-controlled double-blinded randomized clinical trial. Clin Implant Dent Relat Res. 2022 Feb;24(1):116-124. doi: 10.1111/cid.13068. Epub 2022 Jan 24. PMID 35075765